CLINICAL TRIAL: NCT01707823
Title: Prevention of Death From Adenocarcinoma of the Lung by Low Dose Aspirin
Brief Title: Low-Dose Acetylsalicylic Acid in Treating Patients With Stage I-III Non-Small Cell Lung Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Leora Horn, MD, Assistant Professor of Medicine; Assistant Director, Educator Development Program; Clinical Director, Thoracic Oncology Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VICC THN 1227; NCI-2012-01800 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P50CA090949 (NIH)
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Adenocarcinoma of the Lung; Recurrent Non-small Cell Lung Cancer; Stage IA Non-small Cell Lung Cancer; Stage IB Non-small Cell Lung Cancer; Stage IIA Non-small Cell Lung Cancer; Stage IIB Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prevention (acetylsalicylic acid) (Experimental): Patients receive acetylsalicylic acid PO for 7 days.
  Interventions: Drug: acetylsalicylic acid; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: acetylsalicylic acid — Given PO
  Other Names: ASA; Ecotrin; Empirin; Extren
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies low-dose acetylsalicylic acid in treating patients with stage I-III non-small cell lung cancer. Studying samples of urine and blood from patients with cancer in the laboratory may help doctors learn more about changes in biomarkers that occur during treatment with acetylsalicylic acid

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether ASA (acetylsalicylic acid) 325 mg inhibits prostaglandin E2 (PGE2) biosynthesis in patients with early stage non-small cell lung cancer (NSCLC). Cyclooxygenase (COX) catalytic activity will be determined by measuring the metabolite of PGE2, 11alpha-hydroxy-9,12-dioxo-2,3,4,5-tetranor-prostane-1,20 dioic acid (PGE-M) in urine pre- and post-ASA 325 mg as a surrogate of systemic PGE2 biosynthesis.

SECONDARY OBJECTIVES:

I. To determine whether COX-2 protein has a slow turnover in adenocarcinoma of the lung. COX turnover will be determined by measuring urinary PGE-M levels daily for 7 days after discontinuing ASA 325 mg. COX-2 and Prostaglandin expression will also be measured in tumor samples of patients taken at the time of surgery.

OUTLINE:

Patients receive acetylsalicylic acid orally (PO) for 7 days and urine is collected for 7 days post therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have confirmed (stage IIIb-IV) or recurrent non-small cell lung cancer, adenocarcinoma histology
* Understand and voluntarily sign an informed consent document prior to any study related assessments or procedures are conducted
* Anticipated that they will complete all study procedures
* Ability to swallow pills
* No aspirin in the last 7 days

Exclusion Criteria:

* Know allergy to aspirin or other nonsteroidal anti-inflammatory drugs
* History of allergic reaction to aspirin or other non-steroidal anti-inflammatory drugs, including ibuprofen
* Any other concomitant serious illness or organ system dysfunction which in the opinion of the investigator would either compromise patient safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-10; Primary Completion 2018-06 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in PGE2 biosynthesis from baseline and at 14 days after discontinuation of a 7-day course of 325 mg ASA per day | 14 days
  PGE2 is a product of the COX-2 protein. Measurement of its urinary metabolite PGE-M would indicate the level of systemic biosynthesis of PGE2 and thus inhibition of COX-2 product formation.

SECONDARY OUTCOMES:
Change in PGE-M levels from baseline and daily for 7 days after discontinuation of a 7-day course of 325 mg ASA per day | 14 days
  PGE-M is a metabolite of PGE2 in urine. PGE2 is a product of the COX-2 protein. Evidence suggests that COX-2 and PGE2 participate in tumor growth, apoptosis and metastasis, angiogenesis and abrogation of the tumor response. ASA inhibits COX-2. A slow rate of recovery in urinary levels of urinary PGE-M would indicate the rate of catalytically active COX-2 after discontinuation of ASA and may explain the efficacy of once daily low-dose ASA.

CONTACTS AND LOCATIONS:
Overall Officials: Leora Horn, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/